CLINICAL TRIAL: NCT06948565
Title: Prognosis of Cirrhotic Patients Admitted to the General Intensive Care Unit Between 2014 and 2024: a Regional Retrospective Multicentre Cohort Study
Acronym: REACIRRHOSE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/908
Record Dates: First submitted 2025-01-03; First posted 2025-04-29 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-11

CONDITIONS: Cirrhosis; Intensive Care Medicine; Acute on Chronic Liver Failure(ACLF)
Keywords: prognosis; cirrhosis; ICU; ACLF
MeSH Terms: conditions — Fibrosis; Acute-On-Chronic Liver Failure | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational study — This observational study aims to describe the clinical practices and the outcome of patients admitted in ICU.

SUMMARY:
Ten years after our team's publication, practices have changed considerably in the management of severe cirrhotic patients. This study will analyse these practices in primary care hospitals and in a tertiary centre, and assess the impact of these changes on the prognosis of these patients.

The following hypotheses will be tested:

* Improvement in intensive care and overall prognosis compared with data from the literature prior to 2014
* Improved access to liver transplantation compared with the literature prior to 2014
* Improvement in intensive care unit practices (for example: application of recommendations published by learned societies concerning the intensive care unit management of patients with cirrhosis, access to comfort care, degree of clinical severity on admission to the intensive care unit, etc.).
* Centre' effect: variability in the phenotype of patients admitted to intensive care depending on the technical facilities available and whether or not the hospital centre has access to TH.

ELIGIBILITY:
Inclusion Criteria:

Patients with cirrhosis over 18 years of age (cirrhosis either histologically proven or diagnosed by hepatologists according to clinical, biological and ultrasound criteria) admitted to intensive care between January 2014 and December 2024.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cirrhosis admitted to intensive care between January 2014 and December 2024.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
28-day survival | 28 days

SECONDARY OUTCOMES:
Phenotype of patients admitted to intensive care | baseline
Overall survival | through study completion
Survival without liver transplantation | 12 months
Proportion of patients listed for liver transplantation | through study completion
number of patients receiving LT | through study completion
Prognostic performance of general and cirrhosis-specific organ failure scores | baseline
Comparison of the characteristics of patients on admission in primary care hospitals and in university hospital. | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France